CLINICAL TRIAL: NCT04728789
Title: Efficacy and Safety of Avatrombopag in Non-severe Aplastic Anemia - a Multicenter Prospective Single Arm Study
Brief Title: Avatrombopag Usage in NSAA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avatrombopag-1
Record Dates: First submitted 2020-12-01; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Aplastic Anemia; Drug Effect
MeSH Terms: conditions — Anemia, Aplastic | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatrombopag treatment group (Experimental): Avatrombopag would be started with 20mg/day. The dosage would be increased by 20 mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L. The dosage could range from 20mg/week to 60mg/day.
  Interventions: Drug: Avatrombopag 20 MG

INTERVENTIONS:
Drug: Avatrombopag 20 MG — Avatrombopag 20mg/week to 60mg/day, starting at 20mg/day and increased by 20 mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L.

SUMMARY:
This is a multicenter, open-label, prospective one arm study to explore the efficacy and safety of Avatrombopag in non-severe aplastic anemia. Patients meeting the inclusion and exclusion criteria would be recruited. Treatment of Avatrombopag would be started with 20mg/day. The dosage would be increased by 20 mg/day every 2 weeks if the platelet count remains less than 20×10e9/L and reduced if the platelet count reaches over than 150×10e9/L. The dosage could range from 20mg/week to 60mg/day. All patients would receive treatment for at least 6 months except that the platelet <20×10e9/L at the dosage of 60mg/day for 4 weeks or the platelet ≥200×10e9/L at the dosage of 20mg/week for 2 weeks. The hematological response rate and safety will be recorded and compared at every month after starting the study treatment. The patients would be followed up for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed to be non-severe aplastic anemia
2. Patients have at least one of the followings: ①absolute neutrophil count < 1.5×109/L, ②platelet count < 30×109/L, ③ hemoglobin level < 100g/L
3. Patients have no response or relapsed following at least one treatment course in a period time of > 6 months of immunosuppression containing CsA or CsA+anti-thymocyte globulin (ATG);
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
5. Patients able to understand and comply with protocol requirements and instructions and have signed and dated informed consent.

Exclusion Criteria:

1. Congenital aplastic anemia;
2. Presence of chromosomal aberration;
3. Evidence of a clonal hematologic bone marrow disorder (MDS, AML) on cytogenetics;
4. Presence with PNH clone ≥50%;
5. Patients received HSCT before;
6. Uncontrolled infection or bleeding with standard treatment;
7. Allergic to Avatrombopag or accessories;
8. HIV, HCV or HBV active infection or liver cirrhosis or portal hypertension;
9. Patient with QTcF (Fridericia's QT correction formula) at screening <450 msec, or<480 msec with bundle branch block, as determined via the mean of a triplicate ECG and assessed at site, unstable angina pectoris, uncontrolled hypertension(>180/100mmHg)，pulmonary artery hypertension;
10. Have any concomitant malignancies within 5 years expect for local basal cell carcinoma of the skin;
11. Past history of thromboembolic event, heart attack or stroke (including anti-phospholipid antibody syndrome) and current use of anticoagulants;
12. Pregnant or nursing (lactating) woman;
13. Have attended other clinical trials within 3 months;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 Months | 6 months
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR) at 6 months

SECONDARY OUTCOMES:
ORR at 3 Months | 3 months
  ORR will be calculated after 3 months of treatment by measuring platelet, reticulocyte, neutrophil and transfusion independence.
Percentage of patients with clonal evolution at 6 months | 6 months
  Percentage of patients with clonal evolution would be evaluated by bone marrow biopsy at 6 months follow up.
percentage of side effects at 6 months | 6 months
  percentage of side effects would be recorded during the study and be calculated according to CTCAE 5.0 at 6 months
Total volume of Platelet Transfusions | 1 month
  Total volume of Platelet Transfusions
Total volume of Red Blood Cells Transfusions | 1 month
  Total volume of Red Blood Cells Transfusions

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years
Access Criteria: email request

REFERENCES:
- [Derived] Wan Z, Chen M, Han B. Avatrombopag, a promising novel thrombopoietin receptor agonist for refractory/relapsed/intolerant non-severe aplastic anemia: a phase 2 single-arm clinical trial. Ann Med. 2023 Dec;55(1):2224044. doi: 10.1080/07853890.2023.2224044. PMID 37318085